CLINICAL TRIAL: NCT07391085
Title: Augmented Reality Enhances Competency-Based Training in Simulated Vaginal Birth: A Multicenter Randomized Controlled Trial
Brief Title: Augmented Reality Training for Simulated Vaginal Birth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Universidad de Los Andes, Bogota, Colombia (Unknown)
Responsible Party: Principal Investigator, Jorge Carvajal Cabrera, Full Professor of Obstetrics and Gynecology, Pontificia Universidad Catolica de Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB-UC-221212006-2023
Record Dates: First submitted 2026-01-20; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Vaginal Birth Education
Keywords: augmented reality; simulation-based education; vaginal birth; obstetric training; competency-based education; medical education; midwifery education

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned in a parallel design to either a control group receiving conventional text- and video-based preparation or an intervention group receiving the same preparation supplemented with augmented reality-based training. Each participant was exposed to only one study arm.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors were blinded to group allocation. Students were identified only by numeric codes during the simulation, and evaluators completed performance assessments without knowledge of whether participants had received augmented reality training.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Training (Active Comparator): Participants received conventional pre-simulation preparation consisting of text-based materials and an instructional video covering uncomplicated vaginal birth.
  Interventions: Other: Conventional Training
- Augmented Reality Training (Experimental): Participants received conventional text- and video-based preparation supplemented with an augmented reality-based pre-simulation training module.
  Interventions: Other: Augmented Reality Training

INTERVENTIONS:
Other: Conventional Training — Text- and video-based preparation for simulated vaginal birth.
  Arms: Conventional Training
Other: Augmented Reality Training — Augmented reality-based pre-simulation training module for vaginal birth.
  Arms: Augmented Reality Training

SUMMARY:
This study evaluated whether an augmented reality (AR)-based training system improves preparation for simulated vaginal birth compared with traditional text- and video-based learning. Vaginal birth is a complex clinical skill that requires integration of technical actions, situational awareness, and professional behaviors, and opportunities for hands-on training may be limited during undergraduate education.

Undergraduate medical students and midwifery students from two universities in Chile and Colombia were randomly assigned to either conventional preparation (text and instructional video) or the same preparation supplemented with an AR training module. The AR system allowed students to explore a simulated vaginal birth scenario in a self-directed manner before participating in hands-on simulation.

All students then completed a standardized simulated vaginal birth using a high-fidelity simulator as part of their regular curriculum. Performance during the first simulation was assessed by blinded evaluators using a validated Direct Observation of Procedural Skills (DOPS) checklist. The primary outcome was achievement of a predefined minimum competency threshold, with secondary outcomes including overall performance scores, completion of critical tasks, and learner satisfaction.

The goal of this study was to determine whether AR-based pre-simulation training enhances early performance in simulated vaginal birth and could serve as a scalable educational tool to support competency-based training in obstetrics.

DETAILED DESCRIPTION:
This multicenter randomized controlled educational study examined the effectiveness of an augmented reality (AR)-based pre-simulation training system for vaginal birth. The study was conducted at two universities in Chile and Colombia and included undergraduate medical students and midwifery students enrolled in obstetrics and gynecology or women's health courses as part of their regular curriculum.

Participants were randomly assigned to one of two groups. The control group received conventional pre-simulation preparation consisting of written materials and an instructional video covering the management of uncomplicated vaginal birth. The intervention group received the same preparation supplemented with a self-directed AR training module, which allowed learners to explore a simulated vaginal birth scenario, navigate procedural steps, and rehearse task sequencing prior to hands-on simulation.

All participants subsequently completed a standardized simulated vaginal birth using a high-fidelity childbirth simulator. Performance during the first simulation attempt was assessed by blinded evaluators using a previously published and validated Direct Observation of Procedural Skills (DOPS) checklist. The primary outcome was achievement of a predefined minimum competency threshold. Secondary outcomes included overall performance scores, completion of critical tasks, and learner satisfaction with the training experience.

The study was designed to isolate the effect of pre-simulation preparation on initial performance, before learning gains from repeated simulation and debriefing. The findings aim to inform the role of augmented reality as a scalable educational tool to support competency-based training in obstetric education.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate medical students or midwifery students enrolled in obstetrics and gynecology or women's health courses at the participating universities.
* Enrollment in the corresponding academic cohort during the study period.
* Age 18 years or older.
* Willingness to participate and provision of informed consent.

Exclusion Criteria:

* Declined participation or withdrawal of consent.
* Incomplete participation in the simulation session.
* Incomplete or missing performance assessment data.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 389 (Actual)
Dates: Start 2023-03-08 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2024-12-23 (Actual)

PRIMARY OUTCOMES:
Number of participants achieving the minimum competency threshold during simulated vaginal birth | Periprocedural (Day 1, during the first standardized simulated vaginal birth)
  Achievement of a predefined minimum competency threshold assessed using a validated Direct Observation of Procedural Skills (DOPS) checklist during a standardized simulated vaginal birth. Competency was defined as a DOPS score ≥35 with successful completion of all critical items.

SECONDARY OUTCOMES:
Mean Direct Observation of Procedural Skills (DOPS) score during simulated vaginal birth | Periprocedural (Day 1, during the first standardized simulated vaginal birth)
  Overall performance score obtained using the Direct Observation of Procedural Skills (DOPS) checklist (range 0-37), where higher scores indicate better performance, assessed during a standardized simulated vaginal birth.
Number of participants completing all critical tasks during simulated vaginal birth | Periprocedural (Day 1, during the first standardized simulated vaginal birth)
  Successful completion of all predefined critical motor and attitudinal tasks on the DOPS checklist during the first standardized simulated vaginal birth.
Learner satisfaction with the training experience | Immediately after the simulation session
  Participant satisfaction assessed using a post-simulation satisfaction questionnaire on a Likert-type scale (range 1-5), where higher scores indicate greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge A Carvajal, PhD, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Pontificia Universidad Católica de Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to ethical and confidentiality considerations. The dataset includes educational performance assessments of students, collected under informed consent for the purposes of this study only. Data are stored in accordance with institutional policies and applicable regulations, and no plans for public data sharing were approved by the ethics committees.

REFERENCES:
- [Background] Valenzuela, M. T., & Carvajal Cabrera, J. A. (2022). Eficiencia del entrenamiento simulado del parto vaginal en estudiantes de enfermería/obstetricia: The efficiency of simulated vaginal birth training in nursing/midwifery students. ARS MEDICA Revista De Ciencias Médicas, 47(4), 25-31. https://doi.org/10.11565/arsmed.v47i4.1911
- See also: Demonstration video of the augmented reality training module used in the study. — https://vimeo.com/showcase/12060877